CLINICAL TRIAL: NCT04075591
Title: Post-approval Study of Wavefront-guided LASIK for Monovision Treatment of Myopic Subjects With Presbyopia
Brief Title: Wavefront-guided LASIK for Monovision Treatment of Myopic Subjects With Presbyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AMO Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STAR-122-MVPM
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: wavefront-guided LASIK monovision treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Wavefront-guided Lasik Monovision Treatment (Experimental): Wavefront-guided LASIK monovision treatment of myopic subjects with presbyopia using the STAR S4 IR® Excimer laser System with the iDesign Refractive Studio.
  Interventions: Device: iDesign Refractive Studio with STAR S4 IR® Excimer laser System

INTERVENTIONS:
Device: iDesign Refractive Studio with STAR S4 IR® Excimer laser System — Surgeons will perform wavefront-guided monovision LASIK for the treatment of myopic subjects with presbyopia based upon measurements obtained with an iDesign Refractive Studio.

SUMMARY:
This study will be a 12-month, prospective, multicenter, open-label, non-comparative, non-randomized clinical investigation conducted at 8 to 14 sites. A total of 383 subjects will be enrolled to achieve approximately 268 treated subjects, resulting in at least 241 evaluable subjects at the point of refractive stability. After signing the informed consent, subjects meeting all inclusion and exclusion criteria in both eyes may be scheduled for surgery. The follow-up visit schedule will be the same for each operative eye.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and HIPAA authorization.
2. At least 40 years of age at enrollment (date informed consent signed).
3. The refractive error of both subject's eyes, based on the iDesign refraction selected for treatment ("4.0 mm Rx calc" at 12.5 mm), must be myopic with or without astigmatism up to -6.00 D spherical equivalent (SE), with cylinder up to -3.00 D and minimum pre-operative myopia in their non-dominant eye at least as great as their targeted myopic retention.
4. At least one eye must require a myopic treatment.
5. Anticipated stromal bed thickness of at least 250 microns based on preoperative central corneal pachymetry minus the maximum treatment depth to be ablated (as calculated by the iDesign plus the intended flap thickness).
6. Distance Best Spectacle Corrected Visual Acuity (BSCVA) of 20/20 or better.
7. Require an add power of +1.25 D or more but not greater than +2.00 D at 40 cm.
8. Less than or equal to ±0.50 D difference between cycloplegic and manifest refraction sphere.
9. A stable refractive error (based on a previous exam, medical records, lensometry, or prescription that is at least 12 months prior to the preoperative manifest refraction), as defined by a change of less than or equal to

   * 0.50 D in MRSE (sphere and cylinder).
10. Subjects with a history of contact lens wear within the last 4 weeks must discontinue lens wear in order to demonstrate refractive stability according to the following (refractive stability is defined as a change of not more than 0.50 D in manifest refraction sphere and cylinder as well as mean keratometry between measurements): After the Informed Consent process has been completed and subjects are enrolled in the study:

    * Rigid or extended wear contact lenses (toric or spherical) must be removed for at least 3 weeks and soft contact lenses (toric or spherical) for at least 2 weeks prior to the first refraction used to establish stability.
    * After abstaining from contact lens wear for designated time, two consecutive manifest refractions and keratometric readings must be conducted at least 7 days apart
    * I If the subject/eye meets the refractive stability criteria, contact lens wear is not permitted for 2 weeks prior to surgery except as required to test monovision acceptance as described below in the Study Procedures, Contact Lens Trial section NOTE: Refractive stability needs to be confirmed only once during preoperative assessment
11. Agreement between manifest refraction (adjusted for optical infinity) and iDesign System refraction chosen for treatment, as follows:

    * Spherical Equivalent: magnitude of the difference is less than 0.625 D.
    * Cylinder: magnitude of the difference is less than or equal to 0.5 D.
    * Cylinder Axis Tolerance: If either the manifest cylinder entered into the iDesign System or the iDesign cylinder selected for treatment is less than 0.5 D, there is no requirement for axis agreement. When both cylinders have a magnitude of at least 0.5 D, the axis tolerance as determined by the iDesign system is linearly reduced from 15 degrees (0.5 D) to 7.5 degrees (7.0 D) based on the average magnitude of both cylinders. Note: If the axis tolerance is not in the calculated range, the iDesign system will produce a warning and this exam may not be used for treatment planning.
12. Willing and capable of complying with follow-up examinations for the duration of the study.

Exclusion Criteria:

1. Women who are pregnant, breast-feeding, or intend to become pregnant during the study.

   Note: Women who were pregnant or nursing may not be enrolled until 6 months after either delivery or have stopped nursing and there is documented refractive stability.
2. Concurrent use of systemic (including inhaled) medications that may impair healing, including but not limited to: antimetabolites, isotretinoin (Accutane®) within 6 months of treatment, and amiodarone hydrochloride (Cordarone®) within 12 months of treatment. NOTE: The use of inhaled or systemic corticosteroids, whether chronic or acute, within the past 6 months is deemed to adversely affect healing and subjects using such medications are specifically excluded from eligibility.
3. History of any of the following medical conditions, or any other condition that could affect wound healing: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or herpes simplex, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis.

   NOTE: The presence of diabetes (either type 1 or 2), regardless of disease duration, severity, or control, will specifically exclude subjects from eligibility.
4. Subjects with a cardiac pacemaker, implanted defibrillator or other implanted electronic device.
5. History of prior intraocular or corneal surgery (including cataract extraction), active ophthalmic disease or abnormality (including, but not limited to, symptomatic blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization > 1 mm from limbus), retinal detachment/repair, clinically significant lens opacity, clinical evidence of trauma, corneal opacity within the central 9 mm and visible on topography, prior strabismus surgery, strabismus, or at risk for developing strabismus, or with evidence of glaucoma or propensity for narrow angle glaucoma or suspected glaucoma.

   NOTE: Subjects with glaucoma, regardless of medication regimen or control, or an IOP greater than 21 mmHg at screening, are specifically excluded from eligibility.
6. Evidence of keratoconus, corneal dystrophy or irregularity, or abnormal topography.
7. Known sensitivity or inappropriate responsiveness to any of the medications used in the postoperative course.
8. Intolerance to monovision correction based on questionnaire responses to contact lens trial (refer to section Study Procedures, Contact Lens Trial below).
9. Concurrent participation in any other clinical trial, or participation in any other clinical trial within the last 14 days.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
The change in driving scale score from preoperative to postoperative as measured by the driving scale within the PROWL-M (Patient-Reported Outcomes with LASIK for monovision) questionnaire | 12 months
  To assess the effect of monovision LASIK treatment on difficulty with driving as measured by the driving scale within the PROWL-M (Patient-Reported Outcomes with LASIK for monovision) questionnaire
The proportion of subjects who required secondary surgery to reverse monovision | 12 months
  The proportion of subjects who required secondary surgery to reverse monovision will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: AMO Development, LLC Clinical Trial, Study Director — AMO Development, LLC
Locations (10):
- United States (10):
  - Maloney Vision Institute, Los Angeles, California
  - Kraff Eye Institute, Chicago, Illinois
  - Center for Sight, Las Vegas, Nevada
  - Coleman Vision, Albuquerque, New Mexico
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Loden Vision Centers, Goodlettsville, Tennessee
  - Berkeley Eye Institute, P.A., Houston, Texas
  - Texas Eye & Laser Center, Hurst, Texas
  - Utah Eye Center, Ogden, Utah
  - The Eye Center, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu/